CLINICAL TRIAL: NCT06129006
Title: Ultrasound Guided Shoulder Anterior Capsular Infiltration Plus Hydrodilatation With Steroid Versus Hyalase in Patients With Frozen Shoulder
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Yehia Mohamed, principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: frozen shoulder
Record Dates: First submitted 2023-11-08; First posted 2023-11-13 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Frozen Shoulder
MeSH Terms: conditions — Bursitis | interventions — Steroids

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A shoulder anterior capsular infiltration plus hydrodilatation with steroids. (Active Comparator): 25 patients with frozen shoulders treated with ultrasound-guided shoulder anterior capsular infiltration plus hydrodilatation with steroids.
  Interventions: Procedure: hydrodilatation with steroid in group A versus hyalase in group B
- groupB shoulder anterior capsular infiltration plus hydrodilatation with hyalase. (Active Comparator): 25 patients with frozen shoulders treated with ultrasound-guided shoulder anterior capsular infiltration plus hydrodilatation with hyalase.
  Interventions: Procedure: hydrodilatation with steroid in group A versus hyalase in group B

INTERVENTIONS:
Procedure: hydrodilatation with steroid in group A versus hyalase in group B — Hydrodilatation technique:
  the ultrasound transducer will be placed on the posterior surface of the shoulder in the longitudinal plane to identify the posterior glenohumeral joint, bony glenoid, humeral head, and infraspinatus muscle.Then, after sterilizing the area to be injected, the needle will be advanced to the target point between the humeral head cartilage and the infraspinatus tendon using the ultrasound-guided in-plane technique.To ensure the injection into the glenohumeral joint, the Doppler mode will be used to confirm the widening of the space between the humeral cartilage and the innermost synovial line of the infraspinatus muscle by the injected solution.

SUMMARY:
To compare ultrasound-guided shoulder anterior capsular infiltration plus hydrodilatation with a steroid versus hyalase in patients with frozen shoulders

DETAILED DESCRIPTION:
Frozen shoulder (FS) is a self-limiting pathology of the shoulder joint causing restriction in both the active and passive range of movements associated with pain (Konarski et al., 2020).

A frozen shoulder is a common condition causing severe pain and a reduced range of motion in the shoulder. It can result in detrimental effects on quality of life and the ability to perform activities of daily living (ADLs). It affects 2% to 5% of the global population and is more common in diabetic patients. There are a variety of treatment options available for patients with frozen shoulders as part of the management ladder of interventions. FS may persist for more than three years or may never resolve (Sam et al., 2023).

Conservative management includes physiotherapy, NSAIDs, Hydrodilatation (HD), intra-articular steroids, manipulation under anesthesia, and arthroscopic, or open capsular release. Distension of the shoulder capsule with normal saline and steroid infusion has been suggested to benefit by changing the biochemical properties of the capsule in FS (Cho et al., 2019).

Hydrodilatation of the shoulder joint capsule was a novel treatment to alleviate the pain of the affected shoulder. The procedure may be given with or without an adjuvant corticosteroid. Hydrodilatation, using saline and a corticosteroid, was superior in short-term pain reduction and range of motion improvement compared to management using only physiotherapy and corticosteroid injection in patients treated for frozen shoulder (Prasetia et al., 2022).

The proposed hypothesis regarding the mechanism of action in hydrodilatation and pain reduction in patients with frozen shoulder was associated with synovitis and fibrosis removal. Previous studies also noted better pain reduction in patients receiving hydrodilatation with adjuvant corticosteroid than only corticosteroid injection (Albana et al., 2022).

Several other adjuvants were studied in frozen shoulder treatment using hydrodilatation. The hydrodilatation method can cause pain in the shoulder during the intervention, so early manual exercise after the intervention is required to inhibit pain (Wang et al., 2021).

Hyaluronidases are a family of enzymes that catalyze the degradation of hyaluronic acid. By catalyzing the hydrolysis of hyaluronan, a constituent of the extracellular matrix, hyaluronidase lowers the viscosity of hyaluronan, thereby increasing the tissue permeability of injected solutes (Lee et al., 2021).

Accordingly, hyaluronidase is used in medicine in conjunction with other drugs, including steroids, to speed their dispersion and delivery. There is growing evidence that using a steroid in combination with hyaluronidase in shoulder joints or spinal epidural spaces both maximizes the anti-inflammatory properties of the steroid and minimizes the side effects of steroid therapy (Manna et al., 2020).

ELIGIBILITY:
Inclusion Criteria:1- Patients diagnosed with unilateral frozen shoulder. 2- Diagnosis of frozen shoulder will be based on clinical examination (restriction of passive external rotation in the affected shoulder > 50% compared to the opposite side), in the presence of normal plain radiographs (anteroposterior and axillary projections other than calcific tendinopathy).

3- Patients with symptoms for more than three months but less than one year which has not improved with medications and physiotherapy.

4- aged 30 to 70 years old

Exclusion Criteria:

1. History of trauma to the shoulder.
2. History of fracture or dislocation around the shoulder.
3. Inflammatory arthritis
4. coagulation disorders
5. History of previous injections within three months.
6. Cervical radiculopathy.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-11-25 (Estimated); Primary Completion 2025-05-24 (Estimated); Study Completion 2026-12-05 (Estimated)

PRIMARY OUTCOMES:
The Shoulder Pain and Disability Index (SPADI) | baseline and 3 weeks, 3 months, and 12 months after the intervention
  The Shoulder Pain and Disability Index (SPADI) will be used to evaluate pain and disability at baseline and 3 weeks, 3 months, and 12 months after the intervention

REFERENCES:
- [Background] Konarski W, Pobozy T, Hordowicz M, Pobozy K, Domanska J. Current concepts of natural course and in management of frozen shoulder: A clinical overview. Orthop Rev (Pavia). 2021 Jan 28;12(4):8832. doi: 10.4081/or.2020.8832. eCollection 2020 Dec 31. PMID 33585024
- [Background] Sam N, Yusuf I, Idris I, Adnan E, Haryadi RD, Hamid F, Usman MA, Johan MP, Zainuddin AA. A Case Series: Effect of Comorbidities on the Outcomes of Prolotherapy Injection for Frozen Shoulder Patients. Int Med Case Rep J. 2023 Apr 28;16:257-263. doi: 10.2147/IMCRJ.S407723. eCollection 2023. PMID 37143964
- [Background] Cho CH, Bae KC, Kim DH. Treatment Strategy for Frozen Shoulder. Clin Orthop Surg. 2019 Sep;11(3):249-257. doi: 10.4055/cios.2019.11.3.249. Epub 2019 Aug 12. PMID 31475043
- [Background] Prasetia R, Albana R, Herman H, Lesmana R, Chernchujit B, Rasyid HN. Ultrasound-Guided Suprascapular Nerve Block at Spinoglenoid Notch and Glenohumeral Joint Hydrodilation. Arthrosc Tech. 2022 Jun 14;11(7):e1233-e1238. doi: 10.1016/j.eats.2022.03.009. eCollection 2022 Jul. PMID 35936858
- [Background] Albana R, Prasetia R, Primadhi A, Rahim AH, Ismiarto YD, Rasyid HN. The role of suprascapular nerve block in hydrodilatation for frozen shoulder. SICOT J. 2022;8:25. doi: 10.1051/sicotj/2022026. Epub 2022 Jun 14. PMID 35699461
- [Background] Cravioto A, Reyes RE, Ortega R, Fernandez G, Hernandez R, Lopez D. Prospective study of diarrhoeal disease in a cohort of rural Mexican children: incidence and isolated pathogens during the first two years of life. Epidemiol Infect. 1988 Aug;101(1):123-34. doi: 10.1017/s0950268800029289. PMID 3402544
- [Background] Lee JH, Choi EJ, Han SC, Chung HS, Kwon MJ, Jayaram P, Lee W, Lee MY. Therapeutic efficacy of low-dose steroid combined with hyaluronidase in ultrasonography-guided intra-articular injections into the shoulder for adhesive capsulitis. Ultrasonography. 2021 Oct;40(4):555-564. doi: 10.14366/usg.20199. Epub 2021 Feb 22. PMID 34399045